CLINICAL TRIAL: NCT04549532
Title: Multisite Randomized Controlled Trial of Targeted Multidomain (T-MD) Interventions for Complex Mild Traumatic Brain Injury (mTBI)
Brief Title: Targeted Multidomain (T-MD) Interventions for Complex Mild Traumatic Brain Injury (mTBI)
Acronym: T-MD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Inova Health Care Services (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Professor/Research Director, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO20050029; W81XWH2010745 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Concussion, Mild
Keywords: concussion; mTBI
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Design: The current study will employ a single blinded, two-group repeated measures (baseline, 2-week, 4-week, 3-month) design with permuted block random assignment to T-MD and usual care intervention groups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T-MD Intervention Group (Experimental): Participants will be prescribed 1+ interventions tailored to affected domains.Anxiety/Mood-Cog beh therapy(CBT) for maladaptive beliefs/avoidance/coping behaviors. Graded exposure/activity/relaxation exercises, cognitive restructuring. Cognitive-Accommodations for reduced work/school time/delayed deadlines, more frequent/longer cognitive rest during symptom-provoking activities. Migraine/Headache: Education, relaxation training/mindfulness based therapy. Ocular-Exercises for ocular symptoms, near point convergence, may include Brock string, pencil push-ups, fixation, saccade tracking, pursuits. Sleep-Sleep regulation/hygiene. Mindfulness-based training, morning physical activity, CBT.Vestibular-Exercises for dizziness, visual motion sensitivity, gait, imbalance that may include gaze stability, visual habituation, static and dynamic balance/gait.Autonomic-Graded aerobic exercise. Perform daily aerobic exercise, goal 80% HR max on a stationary bike/treadmill/walking/jogging.
  Interventions: Behavioral: Targeted Multidomain
- Behavioral Management (Active Comparator): Participants in control group will receive standardized behavioral management strategies including: activity, hydration, nutrition, sleep, and stress management strategies. These strategies provide general methods to manage concussion symptoms and regulate daily activities to assist in the recovery of concussion. Clinicians will discuss and review a behavioral strategies handout with each participant and answer any questions they may have about the information in the handout. Contact time between clinicians and patients will be similar to avoid effects associated with more or less contact time.
  Interventions: Behavioral: Behavioral Management

INTERVENTIONS:
Behavioral: Targeted Multidomain — Participants in the T-MD intervention group will be prescribed targeted interventions to address each individual's symptoms, impairments, and functional limitations in the areas of anxiety/mood, cognitive, migraine/headache, ocular, vestibular, sleep, autonomic. The length of the intervention period will be 4 weeks or until RTA, whichever comes first.
  Arms: T-MD Intervention Group
Behavioral: Behavioral Management — 1.3. Usual Care (Controls) Group Participants randomized to the usual care (control) group will receive standardized (i.e., all participants in this group will receive the same interventions) behavioral management strategies that include activity, hydration, nutrition, sleep, and stress management strategies.
  Arms: Behavioral Management

SUMMARY:
Objective: This 3-year multisite RCT will determine the effectiveness of a targeted multidomain intervention (T-MD) (anxiety/mood, cognitive, migraine, ocular, vestibular; and sleep, autonomic) compared to usual care (behavioral management) in military-aged civilians with complex mTBI.

DETAILED DESCRIPTION:
A prospective single-blinded two-group multicenter randomized controlled trial (RCT) of a targeted multi-domain intervention in military-aged civilians with complex mTBI will be conducted at the University of Pittsburgh Medical Center Sports Concussion Program (UPitt) and Inova Sports Concussion Clinic. During year 1 the investigators will obtain appropriate contract and research agreements, and institutional, site-specific, and Human Research Protection Official (HRPO) Institutional Review Board (IRB) approvals for the trial. This study will enroll 250 military-aged civilians with a diagnosed complex mTBI from UPitt (125) and Inova (125). Upon enrollment, participants will complete a comprehensive multidomain evaluation of symptoms and impairment that will inform an adjudication process to determine affected clinical profiles and targeted interventions. Participants will then be randomized to either the T-MD or usual care intervention arm. The T-MD group will receive targeted interventions (cognitive behavioral therapy, cognitive accommodations/activities, behavioral regulation for headache/migraine, oculomotor exercises, behavioral sleep intervention, vestibular rehabilitation, graded exertion) for affected clinical profiles based on the adjudication process, whereas usual care will only receive behavioral management strategies (e.g., sleep, nutrition, hydration, activity, stress management). In-clinic treatment sessions will be complemented with at-home activities and compliance will be monitored using a text-based tool. Data collection will include demographic data, medical history, health care utilization (the number of visits and utilization costs), and length of time to return to activity (RTA). Primary outcomes for Aim 1 will be assessed at baseline, 2-week, 4-week, and 3-month post-intervention intervals. Secondary outcomes for Aim 1 will be assessed at baseline, 2-week, and 4-week post-intervention intervals, with select outcomes being measured again at 3-months. The investigators will also determine if participants are recovered (i.e., medically cleared for full return to activity) at 2 weeks, 4 weeks and 3 months post-intervention. Additionally, the investigators will tabulate each participant's healthcare utilization and related costs using electronic health record (EHR) at the conclusion of participation in the study protocol. For Aims 2 and 3, in years 2-3, concurrent measures of brain activation will be obtained (i.e., CBF) in the cerebral cortex using fNIRS for all participants at enrollment and 4 weeks-post intervention. Primary outcome measures for Aims 2 and 3 will be oxygenated (activation) and deoxygenated (deactivation) hemoglobin in regions of interest in the cerebral cortex at rest. Secondary outcomes will include the same fNIRS measures during cognitive and exertion activities. We will control for the time since injury in all analyses. For Aim 1, a linear mixed model will be used to compare primary and secondary outcomes between groups, while accounting for covariates. For Aim 2, a linear mixed model will be used to compare brain regions of interest, while accounting for covariates. For Aim 3, bivariate and partial correlational analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria: Participants must meet ALL of the following inclusion criteria:

* 18-49 years of age
* Normal/corrected vision
* Diagnosed with complex mTBI in the past 8 days-6 months with clear mechanism of injury
* Glascow coma scale (GCS) score no less than 13
* Reported or sign of mTBI including loss of consciousness, amnesia, disorientation/confusion, dizziness, imbalance, memory problems, vomiting
* Complex mTBI-related symptoms and/or impairments in at least one of the following areas: anxiety/mood, cognitive, migraine, ocular, vestibular, sleep, autonomic; per a comprehensive assessment, clinical exam/interview, and adjudication process.

Exclusion Criteria: Participants will be excluded if they meet one or more of the following exclusion criteria:

* History of vestibular disorder (e.g., benign paroxysmal positional vertigo, unilateral, or bilateral vestibular hypofunction)
* History of neurological disorder
* Previous moderate to severe TBI
* History of brain surgery, malformations or tumors
* Diagnosed with cardiac, peripheral or cerebrovascular disease
* Experienced chest pain or shortness of breath while at rest or with mild exertion
* Been told by a doctor to only conduct physical activity under medical supervision
* Previous moderate to severe TBI
* < 8 days or >6 months following current complex mTBI
* Currently pregnant or become pregnant during study
* Currently involved in litigation associated with current or previous mTBI
* Currently on workman's compensation
* Previously participated in the study
* Previously received treatment at either site within last two years as this will unblind treatment group(s)

  * Members of same household will not be included as they may determine their group assignment if more than one person from same household is included and assigned to different groups.

    * Please note that participants with a history of mTBI, ADHD/LD, migraine, or motion sickness will NOT be excluded. We will adjust for any imbalance in the groups on these factors via covariate analysis.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) | NSI will be measured from baseline to 3 months.
  NSI is a 22 item symptom scale, participants will rate the severity of their symptoms on a 5 point likert scale (0, none/rarely ever present to 4, very severe, almost always present). The NSI total score is a sum of the 22 items (range 0-88).
Patient Global Impression of Change (PGIC) | The PGIC will be measured from baseline to 3 months.
  PGIC is a self-reported assessment of change. Participants rate their impression of how much better they feel on a 7 point likert scale. It is a 1 item survey, with higher scores representing no change and associated with feeling worse. (Responses 1=much improved, 2=minimally improved, 3=no change, 4=minimally worse, 5=much worse, 6=very much worse).
Functional Near-infrared Spectroscopy (fNIRS) | fNIRS will be conducted two times, once baseline and again at the 4 week visit.
  fNIRS will be used to record changes in oxygenated hemoglobin (activation) and deoxygenated hemoglobin (deactivation) in participants. fNIRS will assess 3 broad regions of interest: left and right temporal, occipital. It will measure bilateral areas of the inferior frontal, dorsal-lateral prefrontal, and frontal regions of the brain including Brodmann areas as well as the middle frontal gyrus, superior temporal gyrus, and extrastriate visual cortical regions. fNIRS will be done in 2 different paradigms: 1) at rest, and 2) during cognitive activity. At rest measurements will occur while participants are seated, and last about 2 minutes. For the cognitive activity, participants will perform the ImPACT test while wearing the fNIRS unit, and last 20 minutes. We will compare brain activation and deactivation in ROIs across the two points and between rest and cognitive activity paradigms. We will also examine task specific changes within the cognitive test paradigm.

SECONDARY OUTCOMES:
Behavioral Symptom Inventory (BSI-18) | The BSI-18 will be measured from baseline to 3 months.
  The BSI is an 18 item symptom inventory that assesses the level of psychological distress during the past 7 days. Responses are on a 5 point Likert scale (0=not at all - 4 = extremely). The BSI-18 yields total global severity index ranging from 0-72, as well as somatic, depression and anxiety sub-scales. Higher scores indicate higher levels of psychological distress.
Dizziness Handicap Inventory (DHI) | The DHI will be measured from baseline to 3 months.
  The DHI is a 25 item self-reported measure that examines dizziness-related handicap. The assessment has 3 domains (functional, emotional, and physical). Participants self-report the level dizziness has impacted their abilities in the 3 domains with each domain having 9 questions (questions are answered No (0)/Sometimes(2)/Yes(4)) Item scores are summed. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional). Minimum score is 0.
Vestibular Ocular Motor Screening (VOMS) | VOMS will be will be measured from baseline to 4 weeks.
  The VOMS assesses impairment via patient report symptom provocation following each of 5 test components (smooth pursuits, horizontal/vertical saccades, convergence, horizontal and vertical vestibular ocular reflex (VOR) and visual motor sensitivity (VMS). Patients verbally rate changes in headache, dizziness, nausea, and fogginess after each test, as well as report their baseline symptoms. Symptoms in each area are rated on scale 0 (none) to 10 (severe). Scores on any VOMS item of 2+ reflects a positive screening cut-off for vestibular and/or ocular motor impairment.
Modified Balance Error Scoring System (mBESS) | mBESS will be measured from baseline to 4 weeks.
  The mBESS measures postural stability and consists of three stances including feet side by side, a tandem stance, and a single-leg stance on the non-dominant leg. The three stances are performed for 20 seconds each and completed with eyes closed and hand on the iliac crests. Errors include lifting hands off the iliac crests, opening the eyes, stepping, stumbling, or falling, moving the hip into more than a 30 degree of flexion or abduction, lifting the forefoot or heel, or remaining out of the testing position for more than 5 seconds. Each error equals 1 point, with higher scores indicating worse performance. Score ranges from 0-30 (maximum of 10 errors per each stance).
Functional Gait Assessment (FGA) | The FGA will be measured from baseline to 4 weeks.
  FGA is 10 items that assesses the ability of participants to walk with head turns, changes of speed of walking, and walking around obstacles. Each item is scored on a 4 point ordinal scale; 0 (severe impairment), 1 (moderate impairment), 2 (mild impairment), 3 (normal ambulation). Score range is 0-30.
Clinical Profile Screening Inventory (CP Screen) | The CP screen will be measured from baseline to 3 months.
  The CP Screen is a 29 item self-report, clinical profiles based symptom inventory that measures five concussion clinical profiles: 1) anxiety/mood, 2)cognitive/fatigue, 3) migraine, 4) ocular, 5) vestibular; and two modifying factors sleep and cervical. Participants indicate on a scale of 0 (none) to 3 (severe) the level of symptom severity for each item. The CP screen yields an average factor and modifier scores, with higher scores indicative of worse symptom severity, score range is 0-87.
Immediate Post-concussion Assessment and Cognitive Testing (ImPACT) | ImPACT will be administered at baseline, 2 week, 4 week visits.
  ImPACT will be used to assess neurocognitive performance. ImPACT is a computerized neurocognitive test that includes 6 modules: 1) verbal memory, 2) design memory, 3) X's and O's, 4) symbol matching, 5) color matching, and 6) three letter memory. These modules are used to form/score four composite scores - verbal and visual memory 5), visual motor processing speed 6), and reaction time (seconds).
Pittsburgh Sleep Quality Index (PSQI) | The PSQI will be measured from baseline to 3 months.
  The PSQI assesses sleep quality. It is an 19 item self-reported measure that is comprised of seven component scores: 1) subjective sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disturbances, 6) sleep medication usage, and 7) daytime dysfunction. Each item is scored 0-3 (0 = very good, 1 = fairly good, 2= fairly bad, 3=very bad). Higher scores indicate more sleep dysfunction. Score range is 0-21.
Headache Impact Test (HIT-6) | The HIT-6 will be measured from baseline to 3 months.
  The HIT-6 is comprised of 6 self-report items that assess frequency, severity and limitations of daily activities, fatigue, irritability, and concentration related to headaches. Items score from 6 to 13, with higher scores indicating worse severity. Scores = never = 6pts, rarely = 8 pts, sometimes = 10pts, very often = 11 pts, always = 13 points. Score range 36-78.
ID Migraine | ID Migraine will be measured from baseline to 3 months.
  The ID Migraine will be used to screen for headache symptoms. It is a 3 item screening tool designed to assess presence (yes/no) of symptoms related to headache/migraine pain. Scores range from 0-3 with clinical cut-off of 2+ indicating presence of migraines.
Short Form McGill Pain Questionnaire (SF-MPQ) | The SF-MPQ will be measured from baseline to 3 months.
  The SF-MPQ is a 15 item pain scale in which participants rate the intensity of their pain on a 4 point likert scale 0 (none) to 3 (severe). The assessment has two subscales (sensory and affective). Higher scores indicate higher pain. Score range 0-75.
International Physical Activity Questionnaire (IPAQ) | The IPAQ will be measured from baseline to 3 months.
  The International Physical Activity Questionnaire (IPAQ) will be used to assess potential treatment group differences in activity level. The IPAQ is a validated tool to assess recall of average activity level and intensity over the preceding 7 days. Activity levels can be expressed as categorical variables (low, medium, high activity levels) or a continuous variable (MET-minutes/week).
Buffalo Concussion Treadmill Test (BCTT) | The BCTT will be completed at 2 study timepoints (baseline and 4 weeks).
  The BCTT will be used in this study to measure autonomic dysfunction of participants' following mTBI. Prior to test initiation, resting heart rate (HR) is measured after a 2 minute seated resting period. A visual analog scale is used to rate symptoms at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Kontod, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Inova Health System - Inova Sports Medicine Concussion Program, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Per DoD grant requirement, de-identified data will be shared with the Federal Interagency Traumatic Brian Injury Research (FITBIR) informatics system and Congressionally Directed Medical Research Programs (CDMRP).
Time Frame: De-identified data will be shared with FITBIR on an annual basis as required by the funder (DoD).
Access Criteria: Formal requests must be submitted and approved to FITBIR to access this study's de-identified data.
URL: https://fitbir.nih.gov/

REFERENCES:
- [Derived] Zynda AJ, Trbovich AM, Kehinde F, Burley C, Collins MW, Okonkwo DO, Mucha A, Ostop S, Holland C, Perry C, Womble MN, Jennings S, Fedor S, Dollar C, Durfee KJ, Elbin RJ, Kontos AP. Role of anxiety in exercise intolerance and autonomic nervous system dysfunction post-concussion. Neurol Sci. 2025 Aug;46(8):3909-3918. doi: 10.1007/s10072-025-08204-9. Epub 2025 Apr 28. PMID 40293595
- [Derived] Elbin RJ, Trbovich A, Womble MN, Mucha A, Fedor S, Stephenson K, Holland C, Dollar C, Sparto P, Durfee K, Patterson CG, Smith CN, Huppert TJ, Okonkwo DO, Collins MW, Kontos AP. Targeted multidomain intervention for complex mTBI: protocol for a multisite randomized controlled trial in military-age civilians. Front Neurol. 2023 Jun 30;14:1085662. doi: 10.3389/fneur.2023.1085662. eCollection 2023. PMID 37456641